CLINICAL TRIAL: NCT05386732
Title: Safety and Efficacy of the 4MD Microneedling Device in the Treatment of Acne Scars
Brief Title: Safety and Efficacy of the 4MD Micro Needling Device in the Treatment of Acne Scars
Status: Completed | Type: Observational
Sponsor: Dermapenworld (Industry)
Responsible Party: Sponsor
Other Study IDs: Derma_01 1482-N-20
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Acne Scarring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Micro needling — All patients were treated with a 16 needle, 3mm, 33-gauge surgical grade stainless steel needle cartridge. The operator began treatment using a depth of (1mm) and a frequency setting of 4 (corresponding to 120 Hz). Needle depth and frequency was adjusted until pin-point bleeding occured, the minimum and maximum depth used to create pinpoint bleeding was recorded. The operator began treatment using a minimum depth of 1mm and a frequency setting of 4 (corresponding to 120 Hz). Needle depth and frequency was adjusted until pin-point bleeding occurred.

SUMMARY:
The objective of this post market clinical follow-up study is to assess the safety and effectiveness of the 4MD microneedling device in reducing scarring of atrophic acne scars.

The Primary endpoint was to show a reduction in acne scarring in accordance with the Acne Scar Assessment Scale as used by Skinpen (Bellus Medical (DEN160029)).

Goodman and Baron and Jacob acne scar assessment and classification will also be utilized Safety endpoint: incidence of adverse events and side effects

DETAILED DESCRIPTION:
This is a post market study involving 22 healthy patients. Screening data was reviewed to determine eligibility. After informed consent, confidentiality and photographic release forms, participants who meet all inclusion criteria and none of the exclusion criteria were entered into the study. Each patient underwent 2 micro needling sessions 4 weeks apart using the 4MD microneedling device and individual sterile microneedling cartridge (16, 3mm, 33-gauge surgical grade stainless steel needles, arranged in a circular pattern) Patients were assessed at baseline and at week 8. If the assessing physician deemed a 3rd treatment was necessary, the patient underwent the third treatment and would be assessed 4 weeks after the 3rd microneedling treatment Routine VECTRA photography was taken at Baseline, and at the final assessment (4 weeks after what was deemed the last treatment).

Patients' VECTRA photography was used to assess acne scarring at baseline and 4 weeks after the last treatment using the Acne Scar Assessment Scale (DEN160029) by Karnick et al. Assessment was carried out by the principle investigator and 2 blinded physicians.

After each treatment, patients completed a treatment experience assessment and patient diaries including self-assessment of side effects from the day of the treatment to day 7.

The number, type, and severity of adverse events were recorded during the duration of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male & females; 18 to 65 years of age with signs of post-acne facial atrophic scarring.
* Voluntary participation
* Ability to comprehend and provide informed consent.
* Participants agree NOT to use any topical agents containing active ingredients such as retinol, glycolic acid or products that will induce skin peeling or change the appearance of acne scars in the treatment area, during the study period.
* Participants agree NOT to undergo any aesthetic treatments that influence appearing of acne scarring (such as Botox, fillers, microdermabrasion, laser surfacing, chemical peels etc.) in the treatment area, during the study period.
* Participants agree NOT to take part in another clinical study or undergo other treatments during the study period.

Exclusion Criteria:

* Haemophilia / bleeding disorder
* Uncontrolled diabetes mellitus
* Treatment of eyeball or mucosa
* Treatment of skin area with dermatosis, e.g. skin tumor, keloid (or extreme keloidal tendency), solar keratosis, warts, or birth marks
* Anticoagulant therapy, e.g. warfarin, heparin, salicylic acid
* Chemotherapy, radiotherapy, or high doses of corticosteroids
* Systemic infection (e.g. hepatitis) or acute skin infection (e.g. herpes)
* Any form of active acne
* Allergic reaction to topical and local anesthetics
* Pregnancy and lactation
* Eczema, exanthema or open wounds
* Scars not older than 6 months
* Skin area with plastic surgery in the past 12 months
* Skin area with filler or Botox injections in the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male & females; 18 to 65 years of age with signs of post-acne facial atrophic scarring.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Demonstrate a reduction in acne scarring in accordance with the Acne Scar Assessment Scale (DEN160029) 4 weeks after last treatment versus baseline (first treatment). | 4 weeks after last treatment versus baseline (first treatment).
  Demonstrate a reduction in acne scarring in accordance with the Acne Scar Assessment Scale (DEN160029) 4 weeks after last treatment versus baseline (first treatment).
  Scale is a 5 point scale where 0 is no acne scarring and 5 is all or almost all acne scars can be seen with direct lighting.

SECONDARY OUTCOMES:
The time in which redness, pain, and discomfort after treatment decreases. | 4 weeks
  The time in which redness, pain, and discomfort after treatment decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Gabriela Casabona, Marbella, Spain

IPD SHARING:
Plan to Share IPD: No
Data forms part of 510K submission and is confidential